CLINICAL TRIAL: NCT02790788
Title: Physiologic Effects of Stress Dose Corticosteroids in the Management of Inhospital Cardiac Arrest - CORTICA
Brief Title: Physiologic Effects of Steroids in Cardiac Arrest
Acronym: CORTICA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Athens (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, MD, PhD, DEAA, EDIC, Associate Professor of Intensive Care Medicine, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CORTICA-15519/23/5/16
Record Dates: First submitted 2016-05-24; First posted 2016-06-06 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Inhospital Cardiac Arrest
MeSH Terms: interventions — Methylprednisolone; Hydrocortisone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steroids Group (Experimental): Intervention: Stress-dose Steroids. Patients will receive methylprednisolone 40 mg (on the first, postenrollment cardiopulmonary resuscitation cycle. Otherwise, advanced life support will be conducted according to the 2015 guidelines for resuscitation). After resuscitation, patients will be treated with stress-dose hydrocortisone 240 mg daily for 7 days maximum, followed by gradual taper over the next 2 days.
  Interventions: Drug: Methylprednisolone; hydrocortisone
- Control Group (Placebo Comparator): Intervention: Saline placebo. Patients will receive saline placebo on the first, postenrollment cardiopulmonary resuscitation cycle. Otherwise, advanced life support will be conducted according to the 2015 guidelines for resuscitation. After resuscitation, patients will be treated with saline placebo for a maximum of 9 days (i.e. 7 days corresponding to the stress-dose hydrocortisone treatment of the experimental arm plus 2 days corresponding to the gradual taper of the stress-dose hydrocortisone treatment of the experimental arm).
  Interventions: Drug: Saline Placebo

INTERVENTIONS:
Drug: Methylprednisolone; hydrocortisone — Methylprednisolone 40 mg during resuscitation and stress-dose hydrocortisone for postresuscitation shock
  Other Names: Solumedrol; Solucortef
  Arms: Steroids Group
Drug: Saline Placebo — Saline placebo during resuscitation and during the postresuscitation phase.
  Other Names: Isotonic sodium chloride placebo
  Arms: Control Group

SUMMARY:
Early stress-dose steroids are of uncertain efficacy in cardiac arrest. The current authors plan to conduct a prospective, randomized, placebo controlled evaluation of stress-dose steroids efficacy with repect to early postresuscitation hemodynamics, heart function, brain perfusion, and inflammatory response in vasopressor-requiring cardiac arrest. Patients will also be followed for organ dysfunction, potential, steroid-associated complications, and functional outcome at hospital discharge.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Despite recent improvements in the quality of care, in-hospital cardiac arrest is still associated with a high probability of poor outcome. Patients resuscitated from vasopressor-requiring cardiac arrest frequently exhibit early postresuscitation hemodynamic instability that is poorly responsive to hemodynamic support with high vasopressor doses and intravenous fluids titrated to cardiac filling pressures of at least 12 mmHg. Furthermore, preceding studies indicate that postresuscitation disease is a "sepsis-like" syndrome characterized by plasma cytokine elevation, endotoxemia, coagulopathy and adrenal insufficiency contributing to postresuscitation shock. Steroids are currently being used for improving hemodynamics in septic patients, however, their effect on postresuscitation hemodynamics has not been thoroughly elucidated yet.

OBJECTIVES To determine whether stress-dose steroid supplementation during and after cardiopulmonary resuscitation (CPR) improves the hemodynamic parameters (arterial blood pressure, cardiac output, cerebral blood flow) in patients with in-hospital cardiac arrest. Furthermore to study the effects of steroid administration on the inflammatory response and organ failures, and to determine potential, corticosteroid-associated complications such as hyperglycemia, infections, bleeding peptic ulcers and paresis. In summary, we aim to directly assess the physiological effects and safety of steroids during and after CPR. The possible clinical usefulness of steroids during and after CPR - in the context of early postresuscitation hemodynamic support - currently corresponds to an important knowledge gap, as recently acknowledged by Guidelines Evidence Reviewers.

METHODS SETTING Intensive/coronary care units, (ICUs/CCUs) of the Evaggelismos Hospital, Athens, Greece (1,200 beds) and of the Larissa University Hospital, Larissa, Greece (700 beds).

PATIENTS

Inclusion criteria:

Patients who have experienced an in-hospital, vasopressor-requiring cardiac arrest, according to guidelines for resuscitation from 2015.

Exclusion criteria are reported in the dedicated subsection.

ETHICS AND INFORMED CONSENT The study will be conducted in concordance with European Union Clinical Trials Regulation No 536/2014 and the Helsinki Declaration. Due to the emergency situation, consent will not be requested for steroid supplementation during CPR. The patients' families and patients who regain consciousness and communication ability during follow-up will be informed about the study as soon as possible, and any objection will result in exclusion of the patient data from any subsequent analyses. Informed, written next-of-kin consent and non-written patient consent (whenever feasible) will be requested as soon as possible for stress-dose hydrocortisone in postresuscitation shock and continued participation in the study. If consent cannot obtained before patient death, the patient's next of kin will be informed of the study and their permission for inclusion of the patient data in the subsequent analyses will be requested. All consent procedures will additionally be documented on the patient's medical record.

The original protocol version has been approved by the Institutional Review Board (IRB) of Evaggelismos General Hospital on July 14 2016 (Approval No. 126/16-6-2016), and by the IRB of Larissa University Hospital on October 10, 2016 (Approval No. 46113/11-10-2016 - IRB Discussion No. 13/10-10-2016 Θ.6). Subsequent protocol amendments have been approved by the Evaggelismos IRB on January 24, 2017 (Approval No. 8/26-1-2017), and this has been communicated to the IRB of Larissa University Hospital.

STUDY DESIGN We propose a prospective, randomized, double-blind, placebo-controlled, parallel- group clinical trial.

RANDOMIZATION Research Randomizer version 4 (https://www.randomizer.org/) will be used by the study statistician for group allocation. For each study center, random numbers (range, 1-100) will be generated in sets of 4. Each random number of each set will be unique and correspond to 1 of the consecutively enrolled patients. In each set, an odd or even first number will result in assignment of the corresponding patient to the control or steroids group, respectively. In each study center, the group allocation rule will be known solely by the pharmacists who will prepare the study drugs.

CPR AND POSTRESUSCITATION INTERVENTIONS We will enrol adult in-patients with cardiac arrest due to ventricular fibrillation/pulseless tachycardia not responsive to three direct current countershocks, or asystole, or pulseless electrical activity. Study treatments will be administered during the first CPR cycle postenrollment. Patients will be randomized to receive either methylprednisolone 40 mg (Steroids group) or normal saline placebo (Control group) on the first, postenrollment CPR cycle. Otherwise, advanced life support will be conducted according to the 2015 guidelines for resuscitation. After resuscitation, patients will be treated with either stress-dose hydrocortisone of 240 mg daily for 7 days maximum (Steroids group), or saline placebo (Control group). More specifically, at 4 hours after ROSC, patients will receive 100 mL/day (average pump infusion rate ~ 4.2 mL/h) of normal saline that will either contain the stress-dose of hydrocortisone (Steroids group) or solely saline placebo (Control group) for a maximum of 9 days. On days 8 and 9 the hydrocortisone dose of the Steroids group will be tapered to 120 mg and 60 mg, respectively, and finally discontinued on day 10 postrandomization. On ICU/CCU admission, patients will receive a central venous line, and an arterial line, either standard or as part of pulsatility index continuous cardiac output monitoring. Patients with a standard arterial line will also receive a pulmonary artery catheter, provided that attending physicians also agree to this.

DOCUMENTATION AND PATIENT FOLLOW-UP CPR attempts will be documented according to the Utstein style. Hemodynamics and gas-exchange, electrolytes, glucose, central body temperature, lactate and administered fluids and vasopressor/inotropic support will be determined/recorded during CPR, and at ~20 min and ~4 hours as well as at 24, 48 and 72 hours after the return of spontaneous circulation (ROSC); ROSC will be defined as sustained presence of a palpable arterial pulse for at least 20 min. Postresuscitation cardiac output will be monitored for at least 72 hours post-ROSC, and postresuscitation cardiac function will be assessed by ultrasonography within the first hour after ICU admission and at 72 hours post-ROSC. Central-venous blood gas analysis will also be performed at the aforementioned time points and blood samples will be taken for the determination of cytokines at approximately 20 min and 4, 24, 48, and 72 hours post-ROSC.

Follow-up during the first 10 days postrandomization will include 1) Determination/recording of hemodynamics and hemodynamic support, gas-exchange, fluid balance of the preceding 24 hours, and arterial blood lactate and central venous oxygen saturation at 9 a.m.; 2) Daily determinations of serum pro-inflammatory cytokines, and 3) Daily recording (within 8-9 a.m.) of laboratory data, and prescribed medication.

The results of 4 daily determinations (1 every 6 hours) of blood glucose will also be recorded to subsequently analyze the incidence of hyperglycemia (blood glucose exceeding 200 mg/dL -11.1 mmol/L). Follow-up to day 60 post-ROSC will include organ failures, and ventilator-free days. Morbidity/complications throughout ICU/CCU and hospital stay, and times to ICU/CCU and hospital discharge will also be recorded.

Study outcomes are reported in the dedicated subsection.

PROTOCOL AMENDMENTS [Approved, January 24, 2017]

Amendment: 1. Part A: Postresuscitation Cardiac Output (CO) has been moved from the primary to the secondary study outcomes (see also Outcome Measures' subsection). Reason for amendment: We ultimately anticipate to be able to collect such data in <50% of the patients. Part B: Furthermore, the measurement time point of "8 hours postresuscitation" will no longer be part of the protocol and this will apply for the total of the physiological measurements. This aims to limit attending investigator workload.

Amendment 2: Further clarification regarding the "acceptable" time frame for ICU / CCU admission of successfully resuscitated patients. This is a very important logistical issue and will include measures (e.g. monitoring and medical service support and oversight) to optimize the quality of care until ICU admission and the specification of the "maximum acceptable time to ICU admission". In the VSE 1 and 2 studies, this time has been 12 hours. During 2016, the Evaggelismos Department of Intensive Care Medicine has experienced a reduction of 5 ICU beds (i.e. from 30 to 25) and 8 HDU (high-dependency unit) beds from 20 to 12. Therefore, regarding cardiac arrest patients, we have decided to extend the target time limit for admission to 24 hours. Regarding CORTICA, any further delay is to be reported as an "unpreventable" protocol breach, and in the case of a possible extreme circumstance (e.g. a severe flu outbreak), any patients with a projected ICU admission time of more than 48 hours will be excluded. Hence, "a projected ICU admission time of more than 48 hours" will constitute an additional exclusion criterion.

Amendment 3: Further clarification of the "terminal illness" exclusion criterion - life expectancy of no more than 6 weeks): (i) Patients with metastatic cancer [with confirmed bone and/or brain metastases], and/or primary / metastatic disease causing respiratory failure with/without additional organ-system failures [as defined by a corresponding Sequential Organ Dysfunction Assessment (SOFA) subscore of 3 or 4]; (ii) Patients with a pre-arrest worst SOFA score of >=15 (this corresponds to a probability of death of at least 90%); and (ii) Patients with immunosuppression and a new, hospital-acquired septic complication).

Amendment 4: Addition of the following Exclusion Criterion: "Any deviation from the hospital's standard resuscitative procedure" (e.g. poor adherence to the standard Advanced Life Support algorithm such as an epinephrine dosing error or use of atropine, or "unjustified" interruption of chest compressions compromising CPR quality).

Amendment 5: Addition of the following Exclusion Criterion: Pre-arrest diagnosis of an "active" peptic ulcer; that is, either preceding gastroscopic confirmation of a peptic ulcer, or clinical evidence of acute, pre-arrest gastrointestinal bleeding, attributable to peptic ulcer disease.

Amendment 6: Follow-up during the first 10 days: The time of determination of cytokines will be 20 min, 4, 24, 48, and 72 hours post ROSC [as specified in the corresponding outcome measure], and 7 days post-ROSC (that is, the determinations of day 4, 5, 6, 8, 9, and 10 will be cancelled); Reason for change: Study cost reduction.

Amendment 7: An amendment of the statistical analysis plan enabling the inclusion of patients without return of spontaneous circulation (ROSC) was approved by the Evaggelismos Hospital IRB (Approval No. 527/11-11-2021), and by the Larissa University Hospital IRB (Approval No. 44243/10-11-2021. The rationale for this amendment pertained to the prevention of bias due to post-randomization exclusion. The amendment was actually prompted by a relevant peer review comments.

STATISTICS Data will be reported as mean±standard deviation, or median (interquartile range), or number (percentage), unless otherwise specified. Distribution normality will be tested by Kolmogorov-Smirnov test. Dichotomous and categorical variables will be compared by two-sided chi-square or Fisher's exact test. Continuous variables will be compared by two-tailed, independent samples t test or Mann-Whitney exact U test. P- values of multiple t-test comparisons will be subjected to the Bonferroni correction. We will use mixed model analysis to compare repeatedly measured variables between the two groups. Survival data will be analyzed by a previously employed methodology of multivariable Cox regression. Based on previously published data on the mean arterial pressure at 24 hours postresuscitation, to detect an effect size d of 0.761 with an α error probability of 0.015 and power 0.80, we need to enroll a total of 78 patients (39 in each group). A target enrollment of 100 patients with ROSC for at least 20 min will likely adequately compensate for possible dropouts or missing data. Expected results pertain to a steroid-associated benefit with respect to the primary outcomes, consistent with results on secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

Adult in-patients with ROSC [for at least 20 min] after cardiac arrest due to

* Ventricular fibrillation/pulseless tachycardia not responsive to three direct current countershocks, or
* Asystole, or
* Pulseless electrical activity.

Exclusion Criteria:

* Age <18 years
* Terminal illness (i.e. life expectancy <6 weeks e.g. due to metastatic cancer, or Sequential Organ Dysfunction Assessment score of 15 or more, or new septic complication in the presence of immunosuppression) or do-not- resuscitate status
* Cardiac arrest due to exsanguination (e.g. ruptured aortic aneurysm)
* Cardiac arrest before hospital admission
* Pre-arrest treatment with intravenous corticosteroids
* Any history of an allergic reaction
* Transmural myocardial infarction
* Previous enrollment in or exclusion from the current study.
* Confirmation of return of spontaneous circulation before study-drug administration, corresponding to "premature randomization" [reference 18] will also result in patient exclusion due to absence of vasopressor-requiring cardiac arrest.

Additional Exclusion Criteria According to the Protocol Amendment approved on January 24, 2017: Any deviation from the hospital's standard resuscitative procedure.

Pre-arrest diagnosis of an "active" peptic ulcer. Projected ICU admission time of more than 48 hours in case of a concurrent, special public health circumstance (e.g. severe flu outbreak) that may abruptly increase the demand for intensive care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spyros D. Mentzelopoulos, MD, PhD, Principal Investigator — University of Athens; Spyros G. Zakynthinos, MD, PhD, Study Chair — University of Athens
Locations (2):
- Greece (2):
  - Department of Intensive Care Medicine, Evaggelismos Hospital, Athens, Attica
  - Larisa University General Hospital, Larissa, Thessaly

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Girotra S, Nallamothu BK, Spertus JA, Li Y, Krumholz HM, Chan PS; American Heart Association Get with the Guidelines-Resuscitation Investigators. Trends in survival after in-hospital cardiac arrest. N Engl J Med. 2012 Nov 15;367(20):1912-20. doi: 10.1056/NEJMoa1109148. PMID 23150959
- [Background] Al-Alwan A, Ehlenbach WJ, Menon PR, Young MP, Stapleton RD. Cardiopulmonary resuscitation among mechanically ventilated patients. Intensive Care Med. 2014 Apr;40(4):556-63. doi: 10.1007/s00134-014-3247-2. Epub 2014 Feb 26. PMID 24570267
- [Background] Mentzelopoulos SD, Zakynthinos SG, Tzoufi M, Katsios N, Papastylianou A, Gkisioti S, Stathopoulos A, Kollintza A, Stamataki E, Roussos C. Vasopressin, epinephrine, and corticosteroids for in-hospital cardiac arrest. Arch Intern Med. 2009 Jan 12;169(1):15-24. doi: 10.1001/archinternmed.2008.509. PMID 19139319
- [Background] Mentzelopoulos SD, Malachias S, Chamos C, Konstantopoulos D, Ntaidou T, Papastylianou A, Kolliantzaki I, Theodoridi M, Ischaki H, Makris D, Zakynthinos E, Zintzaras E, Sourlas S, Aloizos S, Zakynthinos SG. Vasopressin, steroids, and epinephrine and neurologically favorable survival after in-hospital cardiac arrest: a randomized clinical trial. JAMA. 2013 Jul 17;310(3):270-9. doi: 10.1001/jama.2013.7832. PMID 23860985
- [Background] Adrie C, Adib-Conquy M, Laurent I, Monchi M, Vinsonneau C, Fitting C, Fraisse F, Dinh-Xuan AT, Carli P, Spaulding C, Dhainaut JF, Cavaillon JM. Successful cardiopulmonary resuscitation after cardiac arrest as a "sepsis-like" syndrome. Circulation. 2002 Jul 30;106(5):562-8. doi: 10.1161/01.cir.0000023891.80661.ad. PMID 12147537
- [Background] Adrie C, Laurent I, Monchi M, Cariou A, Dhainaou JF, Spaulding C. Postresuscitation disease after cardiac arrest: a sepsis-like syndrome? Curr Opin Crit Care. 2004 Jun;10(3):208-12. doi: 10.1097/01.ccx.0000126090.06275.fe. PMID 15166838
- [Background] Pene F, Hyvernat H, Mallet V, Cariou A, Carli P, Spaulding C, Dugue MA, Mira JP. Prognostic value of relative adrenal insufficiency after out-of-hospital cardiac arrest. Intensive Care Med. 2005 May;31(5):627-33. doi: 10.1007/s00134-005-2603-7. Epub 2005 Apr 19. PMID 15838680
- [Background] Kim JJ, Lim YS, Shin JH, Yang HJ, Kim JK, Hyun SY, Rhoo I, Hwang SY, Lee G. Relative adrenal insufficiency after cardiac arrest: impact on postresuscitation disease outcome. Am J Emerg Med. 2006 Oct;24(6):684-8. doi: 10.1016/j.ajem.2006.02.017. PMID 16984836
- [Background] Hekimian G, Baugnon T, Thuong M, Monchi M, Dabbane H, Jaby D, Rhaoui A, Laurent I, Moret G, Fraisse F, Adrie C. Cortisol levels and adrenal reserve after successful cardiac arrest resuscitation. Shock. 2004 Aug;22(2):116-9. doi: 10.1097/01.shk.0000132489.79498.c7. PMID 15257083
- [Background] Tsai MS, Huang CH, Chang WT, Chen WJ, Hsu CY, Hsieh CC, Yang CW, Chiang WC, Ma MH, Chen SC. The effect of hydrocortisone on the outcome of out-of-hospital cardiac arrest patients: a pilot study. Am J Emerg Med. 2007 Mar;25(3):318-25. doi: 10.1016/j.ajem.2006.12.007. PMID 17349907
- [Background] Schultz CH, Rivers EP, Feldkamp CS, Goad EG, Smithline HA, Martin GB, Fath JJ, Wortsman J, Nowak RM. A characterization of hypothalamic-pituitary-adrenal axis function during and after human cardiac arrest. Crit Care Med. 1993 Sep;21(9):1339-47. doi: 10.1097/00003246-199309000-00018. PMID 8396524
- [Background] Vaahersalo J, Skrifvars MB, Pulkki K, Stridsberg M, Rosjo H, Hovilehto S, Tiainen M, Varpula T, Pettila V, Ruokonen E; FINNRESUSCI Laboratory Study Group. Admission interleukin-6 is associated with post resuscitation organ dysfunction and predicts long-term neurological outcome after out-of-hospital ventricular fibrillation. Resuscitation. 2014 Nov;85(11):1573-9. doi: 10.1016/j.resuscitation.2014.08.036. Epub 2014 Sep 17. PMID 25238742
- [Background] Bro-Jeppesen J, Kjaergaard J, Stammet P, Wise MP, Hovdenes J, Aneman A, Horn J, Devaux Y, Erlinge D, Gasche Y, Wanscher M, Cronberg T, Friberg H, Wetterslev J, Pellis T, Kuiper M, Nielsen N, Hassager C; TTM-Trial Investigators. Predictive value of interleukin-6 in post-cardiac arrest patients treated with targeted temperature management at 33 degrees C or 36 degrees C. Resuscitation. 2016 Jan;98:1-8. doi: 10.1016/j.resuscitation.2015.10.009. Epub 2015 Oct 23. PMID 26525271
- [Background] Peberdy MA, Andersen LW, Abbate A, Thacker LR, Gaieski D, Abella BS, Grossestreuer AV, Rittenberger JC, Clore J, Ornato J, Cocchi MN, Callaway C, Donnino M; National Post Arrest Research Consortium (NPARC) Investigators. Inflammatory markers following resuscitation from out-of-hospital cardiac arrest-A prospective multicenter observational study. Resuscitation. 2016 Jun;103:117-124. doi: 10.1016/j.resuscitation.2016.01.006. Epub 2016 Jan 27. PMID 26826561
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] Soar J, Nolan JP, Bottiger BW, Perkins GD, Lott C, Carli P, Pellis T, Sandroni C, Skrifvars MB, Smith GB, Sunde K, Deakin CD; Adult advanced life support section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 3. Adult advanced life support. Resuscitation. 2015 Oct;95:100-47. doi: 10.1016/j.resuscitation.2015.07.016. No abstract available. PMID 26477701
- [Background] Link MS, Berkow LC, Kudenchuk PJ, Halperin HR, Hess EP, Moitra VK, Neumar RW, O'Neil BJ, Paxton JH, Silvers SM, White RD, Yannopoulos D, Donnino MW. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S444-64. doi: 10.1161/CIR.0000000000000261. No abstract available. PMID 26472995
- [Background] Fergusson D, Aaron SD, Guyatt G, Hebert P. Post-randomisation exclusions: the intention to treat principle and excluding patients from analysis. BMJ. 2002 Sep 21;325(7365):652-4. doi: 10.1136/bmj.325.7365.652. No abstract available. PMID 12242181
- [Background] REGULATION (EU) No 536/2014 OF THE EUROPEAN PARLIAMENT AND OF THE COUNCIL of 16 April 2014 on clinical trials on medicinal products for human use, and repealing Directive 2001/20/EC. Official Journal of the European Union 2014; L158/1-L158/76.
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Cummins RO, Chamberlain D, Hazinski MF, Nadkarni V, Kloeck W, Kramer E, Becker L, Robertson C, Koster R, Zaritsky A, Bossaert L, Ornato JP, Callanan V, Allen M, Steen P, Connolly B, Sanders A, Idris A, Cobbe S. Recommended guidelines for reviewing, reporting, and conducting research on in-hospital resuscitation: the in-hospital 'Utstein style'. American Heart Association. Circulation. 1997 Apr 15;95(8):2213-39. doi: 10.1161/01.cir.95.8.2213. No abstract available. PMID 9133537
- [Background] Boushel R, Langberg H, Olesen J, Nowak M, Simonsen L, Bulow J, Kjaer M. Regional blood flow during exercise in humans measured by near-infrared spectroscopy and indocyanine green. J Appl Physiol (1985). 2000 Nov;89(5):1868-78. doi: 10.1152/jappl.2000.89.5.1868. PMID 11053338
- [Derived] Mentzelopoulos SD, Pappa E, Malachias S, Vrettou CS, Giannopoulos A, Karlis G, Adamos G, Pantazopoulos I, Megalou A, Louvaris Z, Karavana V, Aggelopoulos E, Agaliotis G, Papadaki M, Baladima A, Lasithiotaki I, Lagiou F, Temperikidis P, Louka A, Asimakos A, Kougias M, Makris D, Zakynthinos E, Xintara M, Papadonta ME, Koutsothymiou A, Zakynthinos SG, Ischaki E. Physiologic effects of stress dose corticosteroids in in-hospital cardiac arrest (CORTICA): A randomized clinical trial. Resusc Plus. 2022 May 26;10:100252. doi: 10.1016/j.resplu.2022.100252. eCollection 2022 Jun. PMID 35652112

RESULTS

PARTICIPANT FLOW:
Groups:
- Steroids Group: Intervention: Stress-dose Steroids. Patients will receive methylprednisolone 40 mg (on the first, postenrollment cardiopulmonary resuscitation cycle. Otherwise, advanced life support will be conducted according to the 2015 guidelines for resuscitation). After resuscitation, patients will be treated with stress-dose hydrocortisone 240 mg daily for 7 days maximum, followed by gradual taper over the next 2 days.
  Methylprednisolone; hydrocortisone: Methylprednisolone 40 mg during resuscitation and stress-dose hydrocortisone for postresuscitation shock
  Of 369 cardiac arrest patients evaluated for eligibility, 100 patients were enrolled of whom 46 were randomized to receive 40 mg of methylprednisolone during resuscitation (first CPR cycle after enrollment), followed by stress dose hydrocortisone, starting at 4 hours postresuscitation in patients with postresuscitation shock.
- Control Group: Intervention: Saline placebo. Patients will receive saline placebo on the first, postenrollment cardiopulmonary resuscitation cycle. Otherwise, advanced life support will be conducted according to the 2015 guidelines for resuscitation. After resuscitation, patients will be treated with saline placebo for a maximum of 9 days (i.e. 7 days corresponding to the stress-dose hydrocortisone treatment of the experimental arm plus 2 days corresponding to the gradual taper of the stress-dose hydrocortisone treatment of the experimental arm).
  Saline Placebo: Saline placebo during resuscitation and during the postresuscitation phase.
  Of 369 cardiac arrest patients evaluated for eligibil ity, 100 patients were enrolled of whom 54 were randomized to receive placebo during resuscitation (first CPR cycle after enrollment), followed by placebo, starting at 4 hours postresuscitation in patients with postresuscitation shock.
Period: Overall Study
Arm/Group | Steroids Group | Control Group
Started | 46 | 54
Completed | 46 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Descriptive Statistics
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroids Group | Control Group | Total
Number analyzed (Participants) | 46 | 54 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.1 (19.2) | 73.2 (12.3) | 72.1 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 44
  Male | 27 | 29 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 46 | 54 | 100
Region of Enrollment [Number; unit: participants]
  Greece | 46 | 54 | 100
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (8.8) | 27.2 (5.9) | 27.4 (7.3)
Hypertension [Count of Participants; unit: Participants] | 31 | 31 | 62
Coronary Artery Disease [Count of Participants; unit: Participants] | 14 | 15 | 29
Diabetes [Count of Participants; unit: Participants] | 14 | 17 | 31
Cardiac Conduction Disturbances [Count of Participants; unit: Participants] | 6 | 7 | 13
Cardiac Arrhythmia [Count of Participants; unit: Participants] | 10 | 15 | 25
Valvular Heart Disease [Count of Participants; unit: Participants] | 8 | 9 | 17
Peripheral Vascular Disease [Count of Participants; unit: Participants] | 8 | 15 | 23
Other Comorbidity [Count of Participants; unit: Participants] | 40 | 42 | 82
Hospital Admission Cause [Medical] [Count of Participants; unit: Participants] | 21 | 36 | 57
Pre-arrest Hospital Stay (days) [Mean (Standard Deviation); unit: Days] | 15.4 (24.6) | 10.6 (17.2) | 12.8 (21.0)
Cardiac Arrest Cause: Hypotension [Count of Participants; unit: Participants] | 29 | 25 | 54
Cardiac Arrest Cause: Myocardial Ischemia [Count of Participants; unit: Participants] | 4 | 4 | 8
Cardiac Arrest Cause: Homeostatic Disorder [Count of Participants; unit: Participants] | 20 | 18 | 38
Cardiac Arrest Cause: Arryhthmia [Count of Participants; unit: Participants] | 9 | 7 | 16
Cardiac Arrest Cause: Other [Count of Participants; unit: Participants] | 3 | 8 | 11
Cardiac Arrest Cause: Respiratory Failure [Count of Participants; unit: Participants] | 29 | 35 | 64

OUTCOME MEASURES:

1. Primary Outcome: Early Postresuscitation Arterial Blood Pressure (mmHg) Measured Through Institution of Invasive Intra-arterial Pressure Monitoring (as Feasible).
Description: Results on early postresuscitation, mean arterial blood pressure (mmHg) are provided for the first, pre-specified time point of measurement, i.e. at 20 min after the return of spontaneous circulation (ROSC).
Time Frame: Time point of measurement: 20 min after the return of spontaneous circulation (ROSC).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 46 | 54
mmHg | 78.4 (21.3) | 75.1 (21.4)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Independent Samples t-test; Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Net) = 3.3, 95% CI 2-sided [-5.2 to 11.8], Standard Error of Mean 4.3

2. Primary Outcome: Early Postresuscitation Central Venous Oxygen Saturation (%) Measured in Blood Samples Obtained Through a Central Venous Catheter Port (as Feasible).
Description: Results on early postresuscitation central venous oxygen saturation (%) are provided for the first, pre-specified time point of measurement, I.e., 20 min after the return of spontaneous circulation (ROSC). Actually, and exclusively for this particular measurement, reasons for the failure of consistent data collection are given below.
Time Frame: Time points of measurement: 20 min after ROSC.
Population: DATA COULD NOT BE COLLECTED; REASON: A CENTRAL VENOUS BLOOD SAMPLE COULD NOT BE CONSISTENTLY OBTAINED AT 20 MIN AFTER RETURN OF SPONTANEOUS CIRCULATION, BECAUSE A CENTRAL VENOUS CATHETER WAS NOT IN PLACE ON MOST OCCASIONS; THE DATA MONITORING COMMITTEE RECOMMENDED THAT THIS SPECIFIC TIME POINT BE EXCLUDED FROM THE ANALYSIS.
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Early Postresuscitation Arterial Blood Pressure (mmHg) Measured Through Institution of Invasive Intra-arterial Pressure Monitoring (as Feasible).
Description: Results on early postresuscitation, mean arterial blood pressure (mmHg) are provided for the second, pre-specified time point of measurement, i.e. at 4 hours after ROSC.
Time Frame: Time points of measurement: 4 hours after ROSC.
Population: DATA COULD NOT BE COLLECTED FROM 7 PATIENTS OF THE STEROIDS GROUP AND FROM 7 PATIENTS OF THE CONTROL GROUP, BECAUSE THESE PATIENTS DIED WITHIN LESS THAN 4 HOURS AFTER ROSC.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 39 | 47
mmHg | 83.9 (18.1) | 78.9 (15.6)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.17, t-test, 2 sided; Mean Difference (Net) = 5.0, 95% CI 2-sided [-2.2 to 12.2], Standard Error of Mean 3.6

4. Primary Outcome: Early Postresuscitation Central Venous Oxygen Saturation (%) Measured in Blood Samples Obtained Through a Central Venous Catheter Port (as Feasible).
Description: Results on postresuscitation central venous oxygen saturation (%) are provided for the second, pre-specified time point of measurement, i.e., at 4 hours after ROSC.
Time Frame: Time points of measurement: 4 hours after ROSC.
Population: DATA COULD NOT BE COLLECTED FROM 17 PATIENTS OF THE STEROIDS GROUP AND FROM 32 PATIENTS OF THE CONTROL GROUP, EITHER BECAUSE PATIENTS DIED WITHIN LESS THAN 4 HOURS AFTER ROSC, OR BECAUSE THEY STILL DID NOT HAVE A CENTRALVENOUS CATHETER IN-PLACE, OR BECAUSE THE ATTENDING INVESTIGATOR DID NOT COLLECT THE REQUIRED CENTRAL VENOUS BLOOD SAMPLE.
Measure: Mean (Standard Deviation); unit: Percent Hemoglobin Concentration
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 29 | 24
Percent Hemoglobin Concentration | 67.4 (10.2) | 56.8 (22.7)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.043, t-test, 2 sided; Mean Difference (Final Values) = 10.6, 95% CI 2-sided [0.4 to 20.8], Standard Error of Mean 5.0

5. Primary Outcome: Early Postresuscitation Arterial Blood Pressure (mmHg) Measured Through Institution of Invasive Intra-arterial Pressure Monitoring.
Description: Results on postresuscitation, mean arterial blood pressure (mmHg) are provided for the third, pre-specified time point of measurement, i.e. at 24 hours after ROSC.
Time Frame: Time points of measurement: 24 hours after ROSC.
Population: DATA COULD NOT BE COLLECTED FROM 11 PATIENTS OF THE STEROIDS GROUP AND FROM 16 PATIENTS OF THE CONTROL GROUP, BECAUSE OF PATIENT DEATH WITHIN LESS THAN 24 HOURS AFTER ROSC.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 35 | 38
mmHg | 79.9 (16.0) | 81.9 (15.2)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.59, t-test, 2 sided; Mean Difference (Net) = -2.0, 95% CI 2-sided [-9.3 to 5.3], Standard Error of Mean 3.7

6. Primary Outcome: Early Postresuscitation Central Venous Oxygen Saturation (%) Measured in Blood Samples Obtained Through a Central Venous Catheter Port.
Description: Results on postresuscitation central venous oxygen saturation (%) are provided for the third, pre-specified time point of measurement, i.e., at 24 hours after ROSC.
Time Frame: Time points of measurement: 24 hours after ROSC.
Population: DATA COULD NOT BE COLLECTED FROM 12 PATIENTS OF THE STEROIDS GROUP AND FROM 20 PATIENTS OF THE CONTROL GROUP, EITHER BECAUSE OF PATIENT DEATH WITHIN LESS THAN 24 HOURS AFTER ROSC, OR BECAUSE THE ATTENDING INVESTIGATOR DID NOT COLLECT THE REQUIRED CENTRAL VENOUS BLOOD SAMPLE.
Measure: Mean (Standard Deviation); unit: Percent Hemoglobin Concentration
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 34 | 34
Percent Hemoglobin Concentration | 71.1 (8.5) | 70.1 (8.3)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.64, t-test, 2 sided; Mean Difference (Net) = 1.0, 95% CI 2-sided [-3.1 to 5.0], Standard Error of Mean 2.0

7. Primary Outcome: Early Postresuscitation Arterial Blood Pressure (mmHg) Measured Through Institution of Invasive Intra-arterial Pressure Monitoring.
Description: Results on postresuscitation, mean arterial blood pressure (mmHg) are provided for the fourth, pre-specified time point of measurement, i.e. at 48 hours after ROSC.
Time Frame: Time points of measurement: 48 hours after ROSC.
Population: DATA COULD NOT BE COLLECTED FROM 17 PATIENTS OF THE STEROIDS GROUP AND FROM 19 PATIENTS OF THE CONTROL GROUP, BECAUSE OF PATIENT DEATH WITHIN LESS THAN 48 HOURS AFTER ROSC.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 29 | 35
mmHg | 80.2 (10.0) | 84.2 (13.6)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.20, t-test, 2 sided; Mean Difference (Net) = -4.0, 95% CI 2-sided [-10.1 to 2.1], Standard Error of Mean 3.0

8. Primary Outcome: Early Postresuscitation Central Venous Oxygen Saturation (%) Measured in Blood Samples Obtained Through a Central Venous Catheter Port.
Description: Results on postresuscitation central venous oxygen saturation (%) are provided for the fourth, pre-specified time point of measurement, i.e., at 48 hours after ROSC.
Time Frame: Time points of measurement: 48 hours after ROSC.
Population: DATA COULD NOT BE COLLECTED FROM 18 PATIENTS OF THE STEROIDS GROUP AND FROM 22 PATIENTS OF THE CONTROL GROUP, EITHER BECAUSE OF PATIENT DEATH WITHIN LESS THAN 24 HOURS AFTER ROSC, OR BECAUSE THE ATTENDING INVESTIGATOR DID NOT COLLECT THE REQUIRED CENTRAL VENOUS BLOOD SAMPLE.
Measure: Mean (Standard Deviation); unit: Percent Hemoglobin Concentration
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 28 | 32
Percent Hemoglobin Concentration | 73.3 (8.0) | 70.5 (6.5)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.14, t-test, 2 sided; Mean Difference (Net) = 2.8, 95% CI 2-sided [-0.9 to 6.6], Standard Error of Mean 1.9

9. Primary Outcome: Early Postresuscitation Arterial Blood Pressure (mmHg) Measured Through Institution of Invasive Intra-arterial Pressure Monitoring.
Description: Results on postresuscitation, mean arterial blood pressure (mmHg) are provided for the fifth, pre-specified time point of measurement, i.e. at 72 hours after ROSC.
Time Frame: Time points of measurement: 72 hours after ROSC.
Population: DATA COULD NOT BE COLLECTED FROM 19 PATIENTS OF THE STEROIDS GROUP AND FROM 20 PATIENTS OF THE CONTROL GROUP, BECAUSE OF PATIENT DEATH WITHIN LESS THAN 72 HOURS AFTER ROSC.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 27 | 34
mmHg | 85.2 (11.6) | 84.7 (14.5)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.90, t-test, 2 sided; Mean Difference (Net) = 0.5, 95% CI 2-sided [-6.4 to 7.3], Standard Error of Mean 3.4

10. Primary Outcome: Early Postresuscitation Central Venous Oxygen Saturation (%) Measured in Blood Samples Obtained Through a Central Venous Catheter Port.
Description: Results on postresuscitation central venous oxygen saturation (%) are provided for the fifth, pre-specified time point of measurement, i.e., at 72 hours after ROSC.
Time Frame: Time points of measurement: 72 hours after ROSC.
Population: DATA COULD NOT BE COLLECTED FROM 19 PATIENTS OF THE STEROIDS GROUP AND FROM 24 PATIENTS OF THE CONTROL GROUP, EITHER BECAUSE OF PATIENT DEATH WITHIN LESS THAN 24 HOURS AFTER ROSC, OR BECAUSE THE ATTENDING INVESTIGATOR DID NOT COLLECT THE REQUIRED CENTRAL VENOUS BLOOD SAMPLE.
Measure: Mean (Standard Deviation); unit: Percent Hemoglobin Saturation
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 27 | 32
Percent Hemoglobin Saturation | 72.5 (9.5) | 70.4 (7.1)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.33, t-test, 2 sided; Mean Difference (Net) = 2.1, 95% CI 2-sided [-2.2 to 6.4], Standard Error of Mean 2.2

11. Secondary Outcome: Left and Right Ventricular Diastolic Area (cm^2) by Echocardiography.
Description: Results are provided on left ventricular end-diastolic area (LVEDA) and right ventricular diastolic area (RVEDA) by echocardiography within 12 hours and 72 hours after ROSC.
Time Frame: Time points of measurement: Within the first 12 hours and at 72 hours postresuscitation.
Population: REASONS FOR MISSING DATA RELATIVE TO TOTAL POPULATION: 1) PATIENT DEATH; 2) NON-ADHERENCE TO PROTOCOL. RVEDA / LVEDA WAS MEASURED AT LEAST ONCE AT 12 / 72 HOURS POST-ROSC IN 42 PATIENTS (20 CONTROL, N=20). FOR EACH ONE OF THE 2 VARIABLES AND TIME POINTS, THE NUMBER OF PATIENTS STUDIED IS =< 22 FOR THE STEROIDS GROUP AND =< 20 FOR THE CONTROL GROUP.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 22 | 20
cm^2
  LVEDA within 12 hours after ROSC: number analyzed (Participants) | 19 | 20
  LVEDA within 12 hours after ROSC | 23.1 (9.1) | 22.8 (8.2)
  RVEDA within 12 hours after ROSC: number analyzed (Participants) | 22 | 19
  RVEDA within 12 hours after ROSC | 12.1 (4.3) | 13.0 (4.0)
  LVEDA at 72 hours after ROSC: number analyzed (Participants) | 15 | 15
  LVEDA at 72 hours after ROSC | 23.1 (7.9) | 18.5 (2.9)
  RVEDA at 72 hours after ROSC: number analyzed (Participants) | 16 | 15
  RVEDA at 72 hours after ROSC | 14.5 (3.7) | 12.6 (4.1)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; REPORTED RESULTS CORRESPOND TO LVEDA WITHIN 12 HOURS AFTER ROSC; Test type: Superiority; p = 0.92, t-test, 2 sided; Mean Difference (Net) = 0.3, 95% CI 2-sided [-5.3 to 5.8], Standard Error of Mean 2.8
Statistical Analysis 2: Comparison: Steroids Group vs Control Group; REPORTED RESULTS CORRESPOND TO RVEDA WITHIN 12 HOURS AFTER ROSC; Test type: Superiority; p = 0.54, t-test, 2 sided; Mean Difference (Net) = -0.81, 95% CI 2-sided [-3.4 to 1.8], Standard Error of Mean 1.3
Statistical Analysis 3: Comparison: Steroids Group vs Control Group; REPORTED RESULTS CORRESPOND TO LVEDA AT 72 HOURS AFTER ROSC; Test type: Superiority; p = 0.048, t-test, 2 sided; Mean Difference (Net) = 4.60, 95% CI 2-sided [0.04 to 9.15], Standard Error of Mean 2.17
Statistical Analysis 4: Comparison: Steroids Group vs Control Group; REPORTED RESULTS CORRESPOND TO RVEDA AT 72 HOURS AFTER ROSC; Test type: Superiority; p = 0.18, t-test, 2 sided; Mean Difference (Net) = 1.9, 95% CI 2-sided [-1.0 to 4.7], Standard Error of Mean 1.4

12. Secondary Outcome: Left and Right Ventricular Ejection Fraction (%) by Echocardiography.
Description: Results are provided on left ventricular ejection fraction (LVEF) and right ventricular ejection fraction (RVEF) within 12 hours and 72 hours after ROSC.
Time Frame: Time points of measurement: Within the first 12 hours and at 72 hours postresuscitation.
Population: Reasons for missing data relative to total population: 1) patient death within 72 hours after ROSC; and 2) non-adherence to protocol. At 72 hours after ROSC, data was not collected from some of the aforementioned patients due to death or because transesophageal echo for the measurement of RVEF was not repeated.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 27 | 29
Percentage
  LVEF within 12 hours after ROSC | 42.3 (14.1) | 45.9 (13.2)
  RVEF within 12 hours after ROSC: number analyzed (Participants) | 19 | 16
  RVEF within 12 hours after ROSC | 41.7 (8.7) | 42.7 (9.3)
  LVEF at 72 hours after ROSC: number analyzed (Participants) | 12 | 14
  LVEF at 72 hours after ROSC | 45 (11.8) | 50 (9.4)
  RVEF at 72 hours after ROSC: number analyzed (Participants) | 12 | 9
  RVEF at 72 hours after ROSC | 42.8 (8.4) | 44.7 (7.1)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; REPORTED RESULTS CORRESPOND TO LVEF WITHIN 12 HOURS AFTER ROSC; Test type: Superiority; p = 0.32, t-test, 2 sided; Mean Difference (Net) = -3.6, 95% CI 2-sided [-10.9 to 3.7], Standard Error of Mean 3.6
Statistical Analysis 2: Comparison: Steroids Group vs Control Group; REPORTED RESULTS CORRESPOND TO RVEF WITHIN 12 HOURS AFTER ROSC; Test type: Superiority; p = 0.76, t-test, 2 sided; Mean Difference (Net) = -1.0, 95% CI 2-sided [-7.2 to 5.3], Standard Error of Mean 3.1
Statistical Analysis 3: Comparison: Steroids Group vs Control Group; REPORTED RESULTS CORRESPOND TO LVEF AT 72 HOURS AFTER ROSC; Test type: Superiority; p = 0.25, t-test, 2 sided; Mean Difference (Net) = -4.9, 95% CI 2-sided [-13.5 to 3.7], Standard Error of Mean 4.2
Statistical Analysis 4: Comparison: Steroids Group vs Control Group; REPORTED RESULTS CORRESPOND TO RVEF WITHIN 72 HOURS AFTER ROSC; Test type: Superiority; p = 0.61, t-test, 2 sided; Mean Difference (Net) = -1.8, 95% CI 2-sided [-9.1 to 5.5], Standard Error of Mean 3.5

13. Secondary Outcome: Eccentricity Index by Echocardiography.
Description: Eccentricity index (ECCI) is defined as the ratio of the left ventricular (LV) "longitudinal" (or anteroposterior) diameter to the LV "transverse" (or septo-lateral) diameter, measured at end diastole and end systole in a short-axis view. Pertinent results are provided for a first determination within 12 hours after ROSC and a second determination at 72 hours after ROSC.
Time Frame: Time points of measurement: Within the first 12 hours and at 72 hours postresuscitation.
Population: Reasons for missing data relative to the total study population were 1) patient death within 72 hours after ROSC; and 2) non-adherence to protocol. Within 12 hours after ROSC, data were obtained from 43 patients (control, n=22). At 72 hours after ROSC, data could not be obtained from all the aforementioned patients, because some of them had died.
Measure: Mean (Standard Deviation); unit: ECCENTRICITY INDEX
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 21 | 22
ECCENTRICITY INDEX
  End-diastolic ECCI within 12 hours after ROSC | 1.2 (0.3) | 1.3 (0.3)
  End-systolic ECCI within 12 hours after ROSC | 1.3 (0.3) | 1.3 (0.3)
  End-diastolic ECCI at 72 hours after ROSC | 1.2 (0.2) | 1.3 (0.3)
  End-systolic ECCI at 72 hours after ROSC | 1.2 (0.3) | 1.3 (0.4)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO END-DIASTOLIC ECCI WITHIN 12 HOURS OF ROSC; Test type: Superiority; p = 0.41, t-test, 2 sided; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.25 to 0.11], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO END-SYSTOLIC ECCI WITHIN 12 HOURS AFTER ROSC; Test type: Superiority; p = 0.38, t-test, 2 sided; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.26 to 0.10], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO END-DIASTOLIC ECCI AT 72 HOURS AFTER ROSC; Test type: Superiority; p = 0.46, t-test, 2 sided; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.29 to 0.14], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO END-SYSTOLIC ECCI AT 72 HOURS AFTER ROSC; Test type: Superiority; p = 0.34, t-test, 2 sided; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.33 to 0.12], Standard Error of Mean 0.11

14. Secondary Outcome: Early Postresuscitation Cardiac Output (L/Min) Measured by Either Pulse Index Continuous Cardiac Output (PiCCO) or a Continuous Cardiac Output (CCO) Thermodilution Pulmonary Artery Catheter.
Description: RESULTS ARE PROVIDED FOR CARDIAC OUTPUT (CO) AT 4 HOURS AFTER ROSC.
Time Frame: Time points of measurement: 4 hours after ROSC.
Population: REASONS FOR MISSING DATA RELATIVE TO TOTAL STUDY POPULATION OF 100: 1) PATIENT DEATH WITHIN 4 HOURS AFTER ROSC; 2) PATIENT STILL NOT IN THE ICU; AND 3) ATTENDING PHYSICIAN OPINION THAT HE/SHE COULD EFFECTIVELY MANAGE THE PATIENT WITHOUT MONITORING OF CO.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 14 | 11
L/min | 4.9 (1.0) | 5.0 (2.0)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.90, t-test, 2 sided; Mean Difference (Net) = -0.10, 95% CI 2-sided [-1.5 to 1.3], Standard Error of Mean 0.65

15. Secondary Outcome: Early Postresuscitation Cardiac Output (L/Min) Measured by Either Pulse Index Continuous Cardiac Output (PiCCO) or a Continuous Cardiac Output (CCO) Thermodilution Pulmonary Artery Catheter.
Description: Results are provided for CO at 24 hours after ROSC.
Time Frame: Time points of measurement: 24 hours after ROSC.
Population: REASONS FOR MISSING DATA RELATIVE TO TOTAL STUDY POPULATION OF 100: 1) PATIENT DEATH WITHIN 24 HOURS AFTER ROSC; 2) PATIENT STILL NOT IN THE ICU; AND 3) ATTENDING PHYSICIAN OPINION THAT HE/SHE COULD EFFECTIVELY MANAGE THE PATIENT WITHOUT MONITORING OF CO.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 26 | 32
L/min | 5.6 (1.6) | 5.4 (1.2)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.59, t-test, 2 sided; Mean Difference (Net) = 0.20, 95% CI 2-sided [-0.54 to 0.94], Standard Error of Mean 0.37

16. Secondary Outcome: Early Postresuscitation Cardiac Output (L/Min) Measured by Either Pulse Index Continuous Cardiac Output (PiCCO) or a Continuous Cardiac Output (CCO) Thermodilution Pulmonary Artery Catheter.
Description: Results are provided for CO at 48 hours after ROSC
Time Frame: Time points of measurement: 48 hours after ROSC.
Population: REASONS FOR MISSING DATA RELATIVE TO TOTAL STUDY POPULATION OF 100: 1) PATIENT DEATH WITHIN 48 HOURS AFTER ROSC; 2) PATIENT STILL NOT IN THE ICU; AND 3) ATTENDING PHYSICIAN OPINION THAT HE/SHE COULD EFFECTIVELY MANAGE THE PATIENT WITHOUT MONITORING OF CO.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 27 | 31
L/min | 5.8 (1.6) | 5.7 (1.3)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.67, t-test, 2 sided; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.60 to 0.93], Standard Error of Mean 0.38

17. Secondary Outcome: Early Postresuscitation Cardiac Output (L/Min) Measured by Either Pulse Index Continuous Cardiac Output (PiCCO) or a Continuous Cardiac Output (CCO) Thermodilution Pulmonary Artery Catheter.
Description: Results are provided for CO at 72 hours after ROSC.
Time Frame: Time points of measurement: 72 hours after ROSC.
Population: REASONS FOR MISSING DATA RELATIVE TO TOTAL STUDY POPULATION OF 100: 1) PATIENT DEATH WITHIN 72 HOURS AFTER ROSC; AND 3) ATTENDING PHYSICIAN OPINION THAT HE/SHE COULD EFFECTIVELY MANAGE THE PATIENT WITHOUT MONITORING OF CO.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 27 | 31
L/min | 5.8 (1.8) | 5.6 (1.3)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.65, t-test, 2 sided; Mean Difference (Net) = 0.19, 95% CI 2-sided [-0.64 to 1.02], Standard Error of Mean 0.41

18. Secondary Outcome: Core Body Temperature in Degrees Celcius.
Description: Results are provided for core body temperature averaged over the following time intervals after ROSC: 1) 0-6 hours; 2) 6-12 hours; 3) 12-18 hours; 4) 18-24 hours; 5) 24-30 hours; 6) 30-36 hours; 7) 36-42 hours; and 42-48 hours.
Time Frame: Time points of measurement: Hourly from intensive care admission to 48 hours postresuscitation.
Population: For the first 6 hours after ROSC, data was collected from 74 patients (Controls, n=40); data was not collected from 26 patients (Controls, n=14), because of "early" death, or "no temperature measurement". For the subsequent time intervals after ROSC, data could not be collected from all the aforementioned 74 patients, because some of them died.
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 34 | 40
Degrees Celcius
  Temperature averaged over 0-6 hours after ROSC | 36.5 (1.1) | 35.6 (5.7)
  Temperature averaged over 6-12 hours after ROSC: number analyzed (Participants) | 33 | 34
  Temperature averaged over 6-12 hours after ROSC | 36.3 (1.0) | 36.6 (1.3)
  Temperature averaged over 12-18 hours after ROSC: number analyzed (Participants) | 33 | 33
  Temperature averaged over 12-18 hours after ROSC | 36.0 (1.0) | 36.5 (1.1)
  Temperature averaged over 18-24 hours after ROSC: number analyzed (Participants) | 33 | 35
  Temperature averaged over 18-24 hours after ROSC | 36.1 (1.5) | 36.3 (0.9)
  Temperature averaged over 24-30 hours after ROSC: number analyzed (Participants) | 32 | 33
  Temperature averaged over 24-30 hours after ROSC | 36.1 (1.1) | 36.2 (1.0)
  Temperature averaged over 30-36 hours after ROSC: number analyzed (Participants) | 31 | 33
  Temperature averaged over 30-36 hours after ROSC | 36.0 (1.1) | 36.2 (1.2)
  Temperature averaged over 36-42 hours after ROSC: number analyzed (Participants) | 31 | 32
  Temperature averaged over 36-42 hours after ROSC | 36.1 (1.0) | 36.2 (1.2)
  Temperature averaged over 42-48 hours after ROSC: number analyzed (Participants) | 31 | 33
  Temperature averaged over 42-48 hours after ROSC | 36.2 (1.0) | 36.3 (1.1)
Statistical Analysis 1: Comparison: Steroids Group; Test type: Superiority; p = 0.41, t-test, 2 sided — RESULTS CORRESPOND TO CORE BODY TEMPERATURE AVERAGED OVER 0-6 HOURS AFTER ROSC; Mean Difference (Net) = 0.8, 95% CI 2-sided [-1.2 to 2.8], Standard Error of Mean 1.0
Statistical Analysis 2: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO CORE BODY TEMPERATURE AVERAGED OVER 12-18 HOURS AFTER ROSC; Test type: Superiority; p = 0.20, t-test, 2 sided; Mean Difference (Net) = -0.36, 95% CI 2-sided [-0.92 to 0.19], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO CORE BODY TEMPERATURE AVERAGED OVER 12-18 HOURS AFTER ROSC; Test type: Superiority; p = 0.07, t-test, 2 sided; Median Difference (Net) = -0.48, 95% CI 2-sided [-1.00 to 0.04], Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO CORE BODY TEMPERATURE AVERAGED OVER 18-24 HOURS AFTER ROSC; Test type: Superiority; p = 0.36, t-test, 2 sided; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.85 to 0.31], Standard Error of Mean 0.29
Statistical Analysis 5: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO CORE BODY TEMPERATURE AVERAGED OVER 24-30 HOURS AFTER ROSC; Test type: Superiority; p = 0.54, t-test, 2 sided; Median Difference (Net) = -0.16, 95% CI 2-sided [-0.66 to 0.35], Standard Error of Mean 0.25
Statistical Analysis 6: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO CORE BODY TEMPERATURE AVERAGED OVER 30-36 HOURS AFTER ROSC; Test type: Superiority; p = 0.62, t-test, 2 sided; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.69 to 0.42], Standard Error of Mean 0.28
Statistical Analysis 7: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO CORE BODY TEMPERATURE AVERAGED OVER 36-42 HOURS AFTER ROSC; Test type: Superiority; p = 0.60, t-test, 2 sided; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.71 to 0.41], Standard Error of Mean 0.28
Statistical Analysis 8: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO CORE BODY TEMPERATURE AVERAGED OVER 42-48 HOURS AFTER ROSC; Test type: Superiority; p = 0.54, t-test, 2 sided; Median Difference (Net) = -0.16, 95% CI 2-sided [-0.69 to 0.36], Standard Error of Mean 0.26

19. Secondary Outcome: Cerebral Blood Flow Index by Near Infrared Spectroscopy With Indocyanine Green.
Description: Results are reported for 2 pairs of cerebral blood flow index (CBFI) measurements performed each time at a lower and a higher level of mean arterial pressure (MAP) at the following time points: 1) at 4 hours after ROSC and 2) at 72 hours after ROSC
Time Frame: Time points of measurement: 4 and 72 hours postresuscitation.
Population: Data were collected from 29 patients (Control, n=15). Reasons for missing data were 1) patient death within less than 72 hours after ROSC; 2) severe postresuscitation shock precluding changes in vasopressor infusion rates to achieve the desired MAP levels; and 3) technical issues with the near infrared spectroscopy equipment.
Measure: Mean (Standard Deviation); unit: nM/s
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 15 | 14
nM/s
  CBFI 4 HOURS POST-ROSC MEAN MAP=75.5 MMHG | 4.0 (2.5) | 3.3 (2.1)
  CBFI 4 HOURS POST-ROSC MEAN MAP=96.0 MMHG | 4.2 (2.3) | 3.5 (1.9)
  CBFI 72 HOURS POST-ROSC MEAN MAP=75.5 MMHG: number analyzed (Participants) | 11 | 14
  CBFI 72 HOURS POST-ROSC MEAN MAP=75.5 MMHG | 4.3 (3.5) | 3.4 (2.2)
  CBFI 72 HOURS POST-ROSC MEAN MAP= 97.0 MMHG: number analyzed (Participants) | 11 | 14
  CBFI 72 HOURS POST-ROSC MEAN MAP= 97.0 MMHG | 4.9 (3.8) | 3.8 (2.4)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO CBFI AT 4 HOURS AFTER ROSC AND AT A MEAN MAP LEVEL OF 75.5 MMHG; Test type: Superiority; p = 0.42, t-test, 2 sided; Mean Difference (Net) = 0.71, 95% CI 2-sided [-2.5 to 1.1], Standard Error of Mean 0.87
Statistical Analysis 2: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO CBFI AT 4 HOURS AFTER ROSC AND AT A MEAN MAP LEVEL OF 96.0 MMHG; Test type: Superiority; p = 0.40, t-test, 2 sided; Median Difference (Net) = 0.68, 95% CI 2-sided [-0.94 to 2.30], Standard Error of Mean 0.79
Statistical Analysis 3: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO CBFI AT 72 HOURS AFTER ROSC AND AT A MEAN MAP LEVEL OF 75.5 MMHG; Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Net) = 0.90, 95% CI 2-sided [-1.49 to 3.28], Standard Error of Mean 1.15
Statistical Analysis 4: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO CBFI AT 72 HOURS AFTER ROSC AND AT A MEAN MAP LEVEL OF 97.0 MMHG; Test type: Superiority; p = 0.36, t-test, 2 sided; Median Difference (Net) = 1.15, 95% CI 2-sided [-1.40 to 3.70], Standard Error of Mean 1.23

20. Secondary Outcome: Organ Failure-free Days.
Description: Number of organ failure-free days during days 1 through 60 postrandomization. Organ failure free=corresponding Sequential Organ Failure Assessment Subscore <3; each subscore can have the following values: 0, 1, 2, 3, and 4; increasing values indicate worsening organ failure.
Time Frame: Days 1 to 60 postrandomization.
Measure: Median (Inter-Quartile Range); unit: Number of Days without Organ Failure
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 46 | 54
Number of Days without Organ Failure | 0 [0 to 13] | 0 [0 to 13]
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.84, Mann Whitney

21. Secondary Outcome: Early Postresuscitation Inflammatory Response as Assessed by Serum Cytokine Levels (pg/mL).
Description: Logarithm (base 10)-transformed serum levels of tumor necrosis factor alpha (TNFa), interleukin (IL)-1 beta, IL-6, IL-8, and IL-10; blood samples were obtained by venipuncture.
Time Frame: Time points of measurement: 4, 24, 48, and 72 hours postresuscitation.
Population: At 4 hours after ROSC, reasons for missing data relative to total study population were 1) patient death within 4 hours after ROSC; and 2) non-adherence to protocol. Regarding the subsequent time points (i.e. 24, 48, and 72 hours), data was collected for <72 patients (Control, n=41), as additional patients died or some samples were not collected.
Measure: Mean (Standard Error); unit: Log(10) transformed values of pg/mL
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 31 | 41
Log(10) transformed values of pg/mL
  IL-6 at 4 hours after ROSC | 2.19 (0.65) | 2.22 (0.57)
  TNFα at 4 hours after ROSC | 1.97 (0.47) | 2.03 (0.47)
  IL-1β at 4 hours after ROSC | 2.07 (0.24) | 2.03 (0.21)
  IL-8 at 4 hours after ROSC | 2.39 (0.36) | 2.43 (0.50)
  IL-10 at 4 hours after ROSC | 1.76 (0.62) | 1.76 (0.76)
  IL-6 at 24 hours after ROSC: number analyzed (Participants) | 26 | 35
  IL-6 at 24 hours after ROSC | 2.06 (0.43) | 1.99 (0.55)
  TNFα at 24 hours after ROSC: number analyzed (Participants) | 27 | 35
  TNFα at 24 hours after ROSC | 2.02 (0.48) | 2.00 (0.51)
  IL-1β at 24 hours after ROSC: number analyzed (Participants) | 27 | 35
  IL-1β at 24 hours after ROSC | 2.06 (0.13) | 2.09 (0.91)
  IL-8 at 24 hours after ROSC: number analyzed (Participants) | 27 | 35
  IL-8 at 24 hours after ROSC | 2.27 (0.41) | 2.29 (0.45)
  IL-10 at 24 hours after ROSC: number analyzed (Participants) | 27 | 35
  IL-10 at 24 hours after ROSC | 1.69 (0.62) | 1.54 (0.65)
  IL-6 at 48 hours after ROSC: number analyzed (Participants) | 21 | 31
  IL-6 at 48 hours after ROSC | 1.87 (0.35) | 1.91 (0.51)
  TNFα at 48 hours after ROSC: number analyzed (Participants) | 21 | 31
  TNFα at 48 hours after ROSC | 1.99 (0.50) | 1.96 (0.50)
  IL-1β at 48 hours after ROSC: number analyzed (Participants) | 21 | 31
  IL-1β at 48 hours after ROSC | 2.09 (0.13) | 2.03 (0.16)
  IL-8 at 48 hours after ROSC: number analyzed (Participants) | 21 | 31
  IL-8 at 48 hours after ROSC | 2.15 (0.37) | 2.17 (0.41)
  IL-10 at 48 hours after ROSC: number analyzed (Participants) | 21 | 31
  IL-10 at 48 hours after ROSC | 1.56 (0.44) | 1.53 (0.44)
  IL-6 at 72 hours after ROSC: number analyzed (Participants) | 24 | 31
  IL-6 at 72 hours after ROSC | 1.93 (0.73) | 1.90 (0.47)
  TNFα at 72 hours after ROSC: number analyzed (Participants) | 24 | 31
  TNFα at 72 hours after ROSC | 2.00 (0.56) | 1.96 (0.51)
  IL-1β at 72 hours after ROSC: number analyzed (Participants) | 24 | 31
  IL-1β at 72 hours after ROSC | 2.05 (0.17) | 2.04 (0.12)
  IL-8 at 72 hours after ROSC: number analyzed (Participants) | 24 | 31
  IL-8 at 72 hours after ROSC | 2.15 (0.38) | 2.19 (0.32)
  IL-10 at 72 hours after ROSC: number analyzed (Participants) | 24 | 31
  IL-10 at 72 hours after ROSC | 1.66 (0.61) | 1.45 (0.48)
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-6 AT 4 HOURS AFTER ROSC; Test type: Superiority; p = 0.86, t-test, 2 sided; Mean Difference (Net) = -0.025, 95% CI 2-sided [-0.311 to 0.262], Standard Error of Mean 0.144
Statistical Analysis 2: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO TNF-α AT 4 HOURS AFTER ROSC; Test type: Superiority; p = 0.56, t-test, 2 sided; Mean Difference (Net) = -0.064, 95% CI 2-sided [-0.287 to 0.158], Standard Error of Mean 0.111
Statistical Analysis 3: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-1β AT 4 HOURS AFTER ROSC; Test type: Superiority; p = 0.52, t-test, 2 sided; Mean Difference (Net) = 0.034, 95% CI 2-sided [-0.071 to 0.139], Standard Error of Mean 0.053
Statistical Analysis 4: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-8 AT 4 HOURS AFTER ROSC; Test type: Superiority; p = 0.70, t-test, 2 sided; Mean Difference (Net) = -0.041, 95% CI 2-sided [-0.254 to 0.172], Standard Error of Mean 0.107
Statistical Analysis 5: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-10 AT 4 HOURS AFTER ROSC; Test type: Superiority; p = 0.97, t-test, 2 sided; Mean Difference (Net) = 0.007, 95% CI 2-sided [-0.326 to 0.340], Standard Error of Mean 0.167
Statistical Analysis 6: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-6 AT 24 HOURS AFTER ROSC; Test type: Superiority; p = 0.61, t-test, 2 sided; Median Difference (Net) = 0.067, 95% CI 2-sided [-0.192 to 0.326], Standard Error of Mean 0.129
Statistical Analysis 7: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO TNFα AT 24 HOURS AFTER ROSC; Test type: Superiority; p = 0.91, t-test, 2 sided; Mean Difference (Net) = 0.014, 95% CI 2-sided [-0.238 to 0.267], Standard Error of Mean 0.126
Statistical Analysis 8: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-1β AT 24 HOURS AFTER ROSC; Test type: Superiority; p = 0.19, t-test, 2 sided; Mean Difference (Net) = -0.040, 95% CI 2-sided [-0.100 to 0.021], Standard Error of Mean 0.030
Statistical Analysis 9: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-8 AT 24 HOURS AFTER ROSC; Test type: Superiority; p = 0.85, t-test, 2 sided; Mean Difference (Net) = -0.022, 95% CI 2-sided [-0.244 to 0.201], Standard Error of Mean 0.111
Statistical Analysis 10: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-10 AT 24 HOURS AFTER ROSC; Test type: Superiority; p = 0.37, t-test, 2 sided; Mean Difference (Net) = 0.147, 95% CI 2-sided [-0.179 to 0.473], Standard Error of Mean 0.162
Statistical Analysis 11: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-6 AT 48 HOURS AFTER ROSC; Test type: Superiority; p = 0.74, t-test, 2 sided; Mean Difference (Net) = -0.043, 95% CI 2-sided [-0.298 to 0.212], Standard Error of Mean 0.127
Statistical Analysis 12: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO ΤΝFα AT 48 HOURS AFTER ROSC; Test type: Superiority; p = 0.80, t-test, 2 sided; Mean Difference (Net) = 0.036, 95% CI 2-sided [-0.246 to 0.318], Standard Error of Mean 0.140
Statistical Analysis 13: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-1β AT 48 HOURS AFTER ROSC; Test type: Superiority; p = 0.20, t-test, 2 sided; Mean Difference (Net) = 0.056, 95% CI 2-sided [-0.030 to 0.142], Standard Error of Mean 0.043
Statistical Analysis 14: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-8 AT 48 HOURS AFTER ROSC; Test type: Superiority; p = 0.83, t-test, 2 sided; Mean Difference (Net) = -0.024, 95% CI 2-sided [-0.246 to 0.198], Standard Error of Mean 0.111
Statistical Analysis 15: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-10 AT 48 HOURS AFTER ROSC; Test type: Superiority; p = 0.83, t-test, 2 sided; Mean Difference (Net) = 0.027, 95% CI 2-sided [-0.223 to 0.276], Standard Error of Mean 0.124
Statistical Analysis 16: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-6 AT 72 HOURS AFTER ROSC; Test type: Superiority; p = 0.85, t-test, 2 sided; Mean Difference (Net) = 0.030, 95% CI 2-sided [-0.294 to 0.354], Standard Error of Mean 0.161
Statistical Analysis 17: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO ΤΝFα AT 72 HOURS AFTER ROSC; Test type: Superiority; p = 0.74, t-test, 2 sided; Mean Difference (Net) = 0.048, 95% CI 2-sided [-0.243 to 0.339], Standard Error of Mean 0.145
Statistical Analysis 18: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-1β AT 72 HOURS AFTER ROSC; Test type: Superiority; p = 0.75, t-test, 2 sided; Median Difference (Net) = 0.013, 95% CI 2-sided [-0.066 to 0.091], Standard Error of Mean 0.039
Statistical Analysis 19: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-8 AT 72 HOURS AFTER ROSC; Test type: Superiority; p = 0.64, t-test, 2 sided; Mean Difference (Net) = -0.045, 95% CI 2-sided [-0.238 to 0.149], Standard Error of Mean 0.096
Statistical Analysis 20: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO IL-10 AT 72 HOURS AFTER ROSC; Test type: Superiority; p = 0.23, t-test, 2 sided; Mean Difference (Net) = 0.179, 95% CI 2-sided [-0.116 to 0.475], Standard Error of Mean 0.147

22. Secondary Outcome: Survival to Hospital Discharge With Favorable Functional Outcome.
Description: Survival to hospital discharge with a Cerebral Performance Category (CPC) Score of 1 or 2. The CPC Score ranges can have the following values: 1, 2, 3, 4, and 5; lower Scores correspond to better outcomes, whereas higher Scores reflect worsening outcomes, e.g. a Score of 4 means Coma or Vegetative state, and a Score of 5 means Brain Death.
Time Frame: Up to 180 days postrandomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 46 | 54
Participants | 2 | 5
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; Test type: Superiority; p = 0.45, Fisher Exact; Percent Difference = 4.9, 95% CI 2-sided [-4.8 to 14.6]

23. Secondary Outcome: Steroid-associated Complications.
Description: Episodes of 1) Hyperglycemia (defined as Blood Glucose >200 mg/dL), 2) Hypernatremia (defined as blood gas analysis-derived sodium ion concentration >150 mEq/L), and 3) Infections (defined as any microbiologically documented, intensive care unit-acquired, or hospital-acquired infection).
Time Frame: Up to 180 days postrandomization.
Measure: Median (Inter-Quartile Range); unit: Number of Episodes per Patient
Arm/Group | Steroids Group | Control Group
Number analyzed (Participants) | 46 | 54
Number of Episodes per Patient
  No. of Episodes of Hyperglycemia | 0 [0 to 2] | 0 [0 to 2]
  No. of Episodes of Hypernatremia | 0 [0 to 0] | 0 [0 to 0]
  No. of Episodes of Infections | 0 [0 to 1] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO THE NUMBER OF EPISODES OF HYPERGLYCEMIA; Test type: Superiority; p = 0.68, Mann Whitney; Mann-Whitney U = 50903.500
Statistical Analysis 2: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO THE NUMBER OF EPISODES OF HYPERNATREMIA; Test type: Superiority; p = 0.68, Mann-Whitney; Mann Whitney U = 52188.5
Statistical Analysis 3: Comparison: Steroids Group vs Control Group; RESULTS CORRESPOND TO THE NUMBER OF EPISODES OF INFECTION; Test type: Superiority; p = 0.37, Mann-Whitney; Mann-Whitney U = 1128.5

ADVERSE EVENTS:
Time Frame: 180 days
Description: Specific Document reporting date of onset of serious adverse event (SAE), SEA location, SAE as unexpected (or not), brief description of affected participant and of SAE, effect of the SAE (e.g. death or life-threatening, etc.), required therapeutic intervention type, relationship of event to study intervention, whether study intervention was discontinued due to the SAE, list of SAE-relevant tests, type of report (initial, follow-up, or final), and list of concurrent medication.
Arm/Group | Steroids Group | Control Group
All-Cause Mortality (participants affected / at risk) | 45/46 | 53/54
Serious Adverse Events (participants affected / at risk) | 45/46 | 53/54
Other Adverse Events (participants affected / at risk) | 23/46 | 33/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steroids Group (N=46) | Control Group (N=54)
Second Cardiac Arrest (General disorders) | 44 (44) | 49 (49) — Second, fatal Cardiac Arrest of various etiologies during follow-up
Cardiac arrest associated multiple organ failure (General disorders) | 19 (19) | 20 (20) — Cardiac arrest associated multiple organ failure causing second cardiac arrest within 72 hours after randomization
Acute Kidney Injury / Renal Failure (General disorders) | 7 (7) | 10 (10) — Acute deterioration in Renal function resulting in a corresponding Sequentiial Organ Dysfunction Assessment sub-score of 3 or more, and/or anuria, and/or need for renal replacement therapy
Severe Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 5 (5) — Drop of platelet count to less than 50000 per microiter
Sepsis / Septic Shock (Infections and infestations) | 18 (18) | 17 (17) — Bacteremia during follow-up, and associated with a systemic inflammatory response, with/without new organ failure(s), with/without need for vasopressors to maintain a mean arterial pressure of 70 mmHg, and with/without lactate exceeding 2.0 mmol/L
Hospital acquired pneumonia (Infections and infestations) | 11 (11) | 9 (9) — New infiltrate in chest x-ray, associated with 1) a systemic inflammatory response, and 2) microbiological evidence from blood and/or bronchial secretions and/or bronchoalveolar lavage
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) — PaO2/FiO2 < 300 mmHg, while ventilated at PEEP of >= 5 cmH2O, bilateral chest x-ray infiltrates, no evidence of cardiogenic pulmonary edema, and patient exposure to a precipitating factor (e.g. aspiration, trauma, etc.) within the last 7 days.
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) — Microbiologically proven infection of the upper urinary tract, associated with a systemic inflammatory response, and/or bacteremia.
Postresuscitation heart failure (General disorders) | 2 (2) | 0 (0) — Postresuscitation cardiac index of less than 2.0 L/min/m2 Body Surface Area requiring inotropic support
New life-threatening arrhythmia (General disorders) | 2 (2) | 3 (3) — New supraventricular or ventricular arrhythmia requiring immediate management according to current Resuscitaiton Guidelines
Hepatic failure (Gastrointestinal disorders) | 0 (0) | 3 (3) — New worsening of liver function associated with a corresponding Sequential Organ Failure Assessment sub-score of 3 or more.
Acute myocardial ischemia (General disorders) | 1 (1) | 2 (2) — New laboratory and electrocardiographic evidence of myocardial ischemia leading to regional dysfunction of the myocardium (e.g. new akinesis/hypokinesis in ultrasound) and requiring a therapeutic intervention.
Paresis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) — Limb and/or respiratory muscle weakness in the context of critical illness associated polyneuropathy / myopathy
Other (General disorders) | 5 (5) | 6 (6) — One case of tension pneumothorax, or status asthmaticus, or gastrointestinal bleeding +/- hemorrhagic shock, or superior vena cava thrombosis, or pancytopenia, or brain edema, or stage IV pressure ulcer, or acute limb ischemia, or pancreatitis.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steroids Group (N=46) | Control Group (N=54)
HYPERGLYCEMIA (General disorders) | 23 (313) | 33 (395) — Number of patients with at least one episode of blood glucose exceeding 200 mg/dL

LIMITATIONS AND CAVEATS:
1. Occurrence of several protocol breaches, with administration of open label steroids to severely shocked patients of both groups
2. Missing central venous oxygen saturation data for the first time point of measurement (i.e. 20 min after ROSC)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-05-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT02790788/Prot_SAP_ICF_003.pdf